CLINICAL TRIAL: NCT03850990
Title: Effect of Gut-Cued Eating on BMI and Efficacy of Open-Label Placebo to Augment Weight Loss
Acronym: GCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mary Boggiano, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300000000
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Eating Behavior; Obesity; Body Weight; Hunger
MeSH Terms: conditions — Feeding Behavior; Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: A single group will be assessed for change in body weight across time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Experimental): In the first visit, this group will learn about placebo pills from a video and will be placebo pills to take twice a day for 8 weeks. They will be asked to take the pills in conjunction with following the weight-loss protocol.
  Interventions: Behavioral: Placebo pill and no placebo pill
- No placebo group (Experimental): In the first visit, this group will learn about placebo pills from a video but will not be given placebo pills. They will follow the weight-loss protocol without placebo pills.
  Interventions: Behavioral: Placebo pill and no placebo pill

INTERVENTIONS:
Behavioral: Placebo pill and no placebo pill — The placebo pills will be green and white gelatin capsules containing microcrystalline cellulose and other inert ingredients.

SUMMARY:
The study will assess the effect of attending to stomach-cues of hunger and fullness on body weight and any additional benefit provided by open-label placebo.

DETAILED DESCRIPTION:
Students and employees from the University of Alabama at Birmingham will consent to four lab visits. On the first visit, they will get measured for a BMI, complete surveys about eating and cognitive styles. They will also get their heart rate and blood pressure taken, and provide a saliva sample for saliva quantification with dental cotton rolls in the mouth before and after a food-craving task (rating computer photos of various foods for liking and desire). They will then see a video explaining the difference between mouth and stomach hunger and instructing them to use a hunger meter to know when to start eating and when to stop eating. They will have a chance to ask questions and will receive a hard copy of the video. They will also receive a satiety tips sheet and will give permission to receive and start receiving daily motivational text messages for the next 2 weeks.

At this time all participants will also watch a short video about placebos and the effect that open-label placebos (non-deceptive placebos; the person knows they are receiving a placebo) have had on previous studies unrelated to obesity or weight loss. If randomized to the placebo group they will take 2 capsules of micro-crystalline cellulose, a non-bioactive ingredient, every day for the duration of the study. Those in the no placebo group will not receive the pills.

The second visit will take place 2 weeks after the first visit. They will be measured for another BMI, complete a meal patterns questionnaire, and have a progress interview about their experience with the new eating instructions. They will receive answers and suggestions corresponding to their interview responses on any challenges faced. Those in the placebo group will have a chance to have any questions or concerns addressed. All participants will then be scheduled for their next visit and will receive the text messages twice a week for the next 3 weeks.

The third visit will take place 3 weeks after the second visit. They will be measured again for a BMI, complete another meal patterns questionnaire, have another progress interview, and get scheduled for their last visit. No text messages will go out between this and the fourth visit.

The fourth visit will take place 3 weeks after the third visit. They will be measured for a BMI and complete another meal patterns questionnaire. They will also get another heart rate, blood pressure, and saliva quantification reading before and after the food-craving task as in the first visit. They will have a final progress interview, followed by a debriefing meeting to let them know more about the study and answer any questions related to any part of the study. They will then be asked if they want to know more about their survey and questionnaire scores. Those in the no placebo group who wish to take placebos will grant permission to be contacted for any future studies that include a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Desire to lose weight
* 18-60 years of age
* Student of employee at the University of Alabama at Birmingham

Exclusion Criteria:

* Current enrollment in commercial weight loss program
* Uncontrolled diabetes
* Uncontrolled hypertension
* Current bipolar disorder
* Current or history of eating disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
BMI | 8 weeks
  Change in body mass index over 8 weeks on the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Boggiano, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- 323 Campbell Hall, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White TR, Wood AS, Ebeling M, Braswell AC, Lausen MA, Isaac S, Gampher JE, Boggiano MM. Change in craving and frequency of consuming palatable foods for non-homeostatic motives after a gut-cued eating intervention. Eat Behav. 2022 Aug;46:101656. doi: 10.1016/j.eatbeh.2022.101656. Epub 2022 Jul 28. PMID 35944376